CLINICAL TRIAL: NCT03063411
Title: Testing a Short Executive Function Training Intervention to Improve Mathematical Reasoning in a Diverse Sample of Children Before They Start School
Brief Title: Testing Whether a Short Training Program Designed to Improve Cognitive Skills Improves 4-year-olds' Maths Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Emma Blakey, Dr, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 146958
Record Dates: First submitted 2017-02-10; First posted 2017-02-24 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cognitive Development
Keywords: Maths reasoning; Working memory; Executive Functions; Cognitive Control; Academic Skills; Randomised Control Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Executive function intervention (Experimental): The intervention comprises four weekly sessions lasting 15-20 minutes. In these sessions, children complete computerised tasks requiring working memory and inhibitory control. These tasks are child friendly and are based on established measures of executive function. The working memory tasks involve maintaining information in mind and processing information (for example, finding items hiding in different locations that move around) and suppressing a dominant but incorrect response (for example, a game where children try to catch fish but not sharks). Children receive feedback on their responses. If children score 75% or more correct in a session the difficulty level increases in the following session.
  Interventions: Other: Executive Function Intervention
- Visual search and simple decision making (Active Comparator): The control task program, like the intervention, comprises four weekly sessions lasting 15-20 minutes. In these sessions, children complete computerised tasks not requiring executive function skills. Instead, they require simple attention and decision making skills and visual search skills. For example, finding an item among distractors (e.g., a spaceship), or deciding which of two animals can fly (out of a bird and a fish). Children receive feedback on their responses.
  Interventions: Other: Active Control Group

INTERVENTIONS:
Other: Executive Function Intervention — In the executive function training group, children will complete computerised tasks requiring working memory and inhibitory control over four weekly sessions lasting 15-20 minutes. The aim is to improve their executive function skills. In the active control group, children will complete computerised tasks requiring simple decision making and visual search skills over four weekly sessions lasting 15-20 minutes.
  Arms: Executive function intervention
Other: Active Control Group — This is the active control condition. Children will complete computerised tasks requiring simple decision making and visual search skills over four weekly sessions lasting 15-20 minutes.
  Arms: Visual search and simple decision making

SUMMARY:
This study will test whether a short training program - designed to improve memory and attention skills - will benefit mathematical reasoning in preschoolers from a range of socio-economic backgrounds. The investigators will test how long any benefits last for and whether any intervention effects are greater for children from disadvantaged backgrounds. The aim is to test interventions that aim to close the achievement gap by improving skills known to underpin academic skills, at an age children may benefit most from training.

DETAILED DESCRIPTION:
Children's academic success across a range of domains is related to their executive function skills - specifically by their ability to maintain and update information (working memory) and to suppress inappropriate responses (inhibitory control). These skills undergo significant development during the preschool years. Notably, preschool executive function skills strongly predict school readiness, as well as concurrent and later academic achievements in mathematics. The aim of this project is to test an intervention that is specifically designed to improve preschoolers' executive functions - crucially, before the achievement gap sets in. The study will be carried out, following CONSORT (2010) guidelines, with typically developing preschoolers (aged approximately 4 years of age). The study will include children from socioeconomically advantaged and disadvantaged families. Children will be randomly assigned to either an executive function training group or an active control group. A nominated person external to the project will conduct the random allocation process. The random allocation will be done for each nursery to ensure roughly even numbers in each group from each nursery. Children in both groups will complete computerized tasks lasting 15-20 minutes once a week for four weeks. The investigators will compare the trained children to an active control group that closely matches the training in terms of activity. To check for improvements, the investigators will measure cognitive and maths skills at baseline (one week before training); one week post-training; three months post-training; and one year post-training. These assessments will be conducted by testers blind to the child's group.

ELIGIBILITY:
Inclusion criteria:

* Must be attending a nursery school attached to a primary school.
* Must speak and understand English (class teachers will advise on this).
* Must have at least one measure of working memory completed at baseline and one measure of inhibitory control completed at baseline.

Exclusion criteria:

* Must not have a significant diagnosed or known physical, mental or learning disability.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in mathematical reasoning scores as measured by the WIAT-II mathematical reasoning sub-test. | Baseline = one week before the intervention; post-test = one week post-intervention, three months post-intervention.
  The investigators will use the Wechsler Individual Achievement Test-II to measure this (WIAT-II; Wechsler, 2005).

SECONDARY OUTCOMES:
Long-term change in mathematical reasoning as measured by the WIAT-II mathematical reasoning sub-test. | One year post-training from baseline
Change in verbal working memory as measured by the Backward Word Span task. | One week post-intervention from baseline, three months post-intervention from baseline and 1 year post-intervention from baseline.
Change in visuo-spatial working memory as measured by the Corsi Block task. | One week post-intervention from baseline, three months post-intervention from baseline and 1 year post-intervention from baseline.
Change in in inhibitory control as measured by the Grass/Snow task. | One week post-intervention from baseline, three months post-intervention from baseline and 1 year post-intervention from baseline.
Change in in inhibitory control as measured by the Peg Tapping task. | One week post-intervention from baseline, three months post-intervention from baseline and 1 year post-intervention from baseline.
Change in classroom engagement score as rated by teachers using the Classroom Engagement Scale (FitzPatrick & Pagani, 2012). | Three months post-intervention from baseline and 1 year post-intervention from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Our Funder: The Nuffield Foundation — http://www.nuffieldfoundation.org/trialling-executive-function-training-intervention-preschoolers